CLINICAL TRIAL: NCT03437642
Title: Retrospective and Prospective Observational Study on Cardiological and Oncological Psychosomatics
Brief Title: Psyhosomatic Medicine in Oncologic and Cardiac Disease Study
Acronym: PSYCHONIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: San Filippo Neri General Hospital (Other)
Responsible Party: Principal Investigator, Christian Pristipino, MD, Head of Research and Training section, Interventional Cardiology Unit, San Filippo Neri General Hospital
Other Study IDs: v24-9-2017
Record Dates: First submitted 2017-12-22; First posted 2018-02-19 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Acute Myocardial Infarction; Tako Tsubo Cardiomyopathy; Breast Cancer
MeSH Terms: conditions — Takotsubo Cardiomyopathy; Breast Neoplasms | interventions — Psychotherapy, Brief

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Tako-Tsubo - STP: Short term psychotherapy + Classic cardiological therapy
  Interventions: Behavioral: Short Term Psychotherapy
- Tako-Tsubo - Control: Classic cardiological therapy only
- Oncologic - STP: Short term psychotherapy + Classic oncological therapy
  Interventions: Behavioral: Short Term Psychotherapy
- Oncologic - Control: Classic oncological therapy only
- AMI - STP: Short term psychotherapy + Classic cardiological therapy
  Interventions: Behavioral: Short Term Psychotherapy
- AMI - Control: Classic cardiological therapy only
- Healthy Subjects: No therapy

INTERVENTIONS:
Behavioral: Short Term Psychotherapy — Humanistic-existential psychotherapy derived from ontopsychological method and specifically adapted to public health systems. Individual and group sessions to be tailored to individual needs
  Groups: AMI - STP; Oncologic - STP; Tako-Tsubo - STP

SUMMARY:
Psychological processes play a complex role in the pathophysiology of many diseases. However, the body and emotional perception of patients and the relationship between dreams and disease still need to be investigated.

The investigators planned an observational and controlled research aimed at assessing some previously unaddressed baseline psychological characteristics and their changes at 1 and 5 years after a short-term psychotherapy in carefully characterised patients with heart or oncologic diseases .

The patients that will be enrolled are:

* 50 patients ≤ 75 year old with acute myocardial infarction;
* 30 patients ≤ 75 year old with Tako-Tsubo syndrome;
* 50 women ≤ 75 year old, recently operated on breast cancer:
* 90 control subjects of the same age and gender of the enrolled patients, without relevant pathologies during the last 10 years. Relevant pathologies are defined as those that required a hospitalisation or a long-lasting medical therapy.

At the enrolment all the subjects will undergo a complete medical evaluation, and the following psychometric tests: Self-evaluation test, Social Support Questionnaire, Beck Depression Inventory II (BDI II), MacNew Heart Disease Health-Related Quality of Life Questionnaire, State-Trait Anxiety Inventory (STAI), State-Trait Anger Expression Inventory (STAXI 2).

In two distinct following meetings, an open questionnaire exploring the body and emotional perception, and another exploring past and recent dreams, will be administered.

The same evaluation will be done for the healthy subjects.

After the initial evaluation, all the patients will be given the choice to start a short-term psychotherapy lasting 6 months on top of medical therapy or to continue classic medical therapy only. Healthy subjects will be not offered the possibility to follow psychotherapy.

At first year of follow-up, the battery of psychometric test, and the two questionnaires exploring the body and emotional perception, and changes and characteristics of dreams during the psychotherapy, will be re-administered.

The following data will be evaluated:

Psychological characteristics at follow-up. Incidence of new relevant medical events Quality of life Relationship between psychological characteristics and health status, and quality of life

At 5 year follow-up psychometric tests and the clinical data will be evaluated in all the groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients within one week from an Acute myocardial infarction treated with primary or urgent PCI
* Patients within one week from the onset of Tako Tsubo cardiomyopathy.
* Patients with a diagnosis of breast cancer in the preceding six months
* Age and sex matched control subjects without relevant medical pathologies in the preceding 10 years

Exclusion Criteria:

* Cognitive impairment
* Refusing the enrolment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * 50 patients ≤ 75 year old with acute myocardial infarction;
  * 30 patients ≤ 75 year old with Tako-Tsubo syndrome;
  * 50 women ≤ 75 year old, recently operated on breast cancer:
  * 90 control subjects of the same age and gender of the enrolled patients, without relevant pathologies during the last 10 years. Relevant pathologies are defined as those that required a hospitalisation or a long-lasting medical therapy.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2018-03-27 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of new relevant medical events | at 1 year
  Relevant medical events are defined as any new medical condition significantly impairing normal daily activities or requiring hospitalization or needing specific and permanent drug treatment.

SECONDARY OUTCOMES:
Cumulative incidence of new relevant medical events | at 5 years
  Relevant medical events are defined as any new medical condition significantly impairing normal daily activities or requiring hospitalization or needing specific and permanent drug treatment.
Changes in body perception and dreams | at 1 year
  These changes will be evaluated with dedicated qualitative questionnaires formulated with open questions.
Incidence of rehospitalisations | at 1 year
  Number of rehospitalisations during the first year of follow-up
Incidence of rehospitalisations | at 5 years
  Number of rehospitalisations during 5 years follow-up
Distress grade | at 1 year
  Self-evaluation test (score range 1-10, higher stress for higher values)
Distress grade | at 5 years
  Self-evaluation test (score range 1-10, higher stress for higher values)
Depression symptoms | at 1 year
  Beck depression inventory II (score range 0-63, more severe depression symptoms for higher values)
Depression symptoms | at 5 years
  Beck depression inventory II (score range 0-63, more severe depression symptoms for higher values)
Social support | at 1 year
  Social support questionnaire (score range 12-72, the higher the score the lower the support)
Social support | at 5 year
  Social support questionnaire (score range 12-72, the higher the score the lower the support)
Quality of life | at 1 year
  Mac New Health-related quality of life questionnaire (score range 1-7, the higher the score the higher the quality of life, 4 subscales not merged)
Quality of life | at 5 years
  Mac New Health-related quality of life questionnaire (score range 1-7, the higher the score the higher the quality of life, 4 subscales not merged)
Anxiety grade | At 1 year
  State-Trait Anxiety inventory (score range 20-80, the higher the score the more anxiety the patients has, 2 subscales)
Anxiety grade | At 5 years
  State-Trait Anxiety inventory (score range 20-80, the higher the score the more anxiety the patients has, 2 subscales)
Anger level | at 1 year
  State-Trait Anger Expression inventory (score range 0%-100%, the higher the score the higher the anger, two subscales)
Anger level | at 5 years
  State-Trait Anger Expression inventory (score range 0%-100%, the higher the score the higher the anger, two subscales)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Roncella, MD, Principal Investigator — San Filippo Neri General Hospital
Locations (1):
- San Filippo Neri General Hospital, Roma, Italy

REFERENCES:
- [Derived] Roncella A, Pristipino C, Di Carlo O, Ansuini M, Corbosiero A, Di Fusco SA, Palumbo G, Gigantesco A, Mirabella F, De Angelis R, Pasceri V, Cancellara L, Colivicchi F, Allan R, Mirri MA, Speciale G. PSYChosomatic Medicine in ONcologIc and Cardiac Disease (PSYCHONIC) Study-A Retrospective and Prospective Observational Research Protocol. J Clin Med. 2021 Dec 10;10(24):5786. doi: 10.3390/jcm10245786. PMID 34945081